CLINICAL TRIAL: NCT01509768
Title: An Observational Prospective Natural History Study of Patients With Mucopolysaccharidosis Type IIIB (MPS IIIB, Sanfilippo Syndrome Type B)
Brief Title: Natural History Study of Patients With Mucopolysaccharidosis Type IIIB (MPS IIIB, Sanfilippo Syndrome Type B)
Status: Completed | Type: Observational
Sponsor: Shire (Industry)
Responsible Party: Sponsor
Organization: Takeda (Industry)
Other Study IDs: HGT-SNB-088
Record Dates: First submitted 2012-01-10; First posted 2012-01-13 (Estimated); Last update posted 2021-03-17 (Actual); Status verified 2021-03

CONDITIONS: Sanfilippo Syndrome Type B
Keywords: MPS IIIB
MeSH Terms: conditions — Mucopolysaccharidosis III

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — blood (plasma and serum), cerebrospinal fluid (CSF), urine
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- No treatment: This is a longitudinal, prospective, observational, natural history study of patients with MPS IIIB to identify endpoints that may be used for future ERT trials via standardized clinical, biochemical, neurocognitive, developmental, behavioral and imaging measures

SUMMARY:
The purpose of this study is to evaluate the natural course of disease progression in Mucopolysaccharidosis Type III (MPS IIIB) patients who are untreated to identify potential surrogate endpoints that may be utilized in future treatment trials of MPS IIIB using predefined assessments including standardized clinical, biochemical, neurocognitive, developmental, and imaging measures.

DETAILED DESCRIPTION:
This is a multicenter longitudinal, prospective, natural history study of patients with MPSIIIB designed to identify potential surrogate endpoints that may be utilized in future Enzyme replacement therapy (ERT) trials of MPS IIIB via defined assessments including standardized clinical, biochemical, neurocognitive, development, and imaging measures.

ELIGIBILITY:
Inclusion Criteria:

Each patient must meet all of the following criteria to be enrolled in this study.

1. Definitive diagnosis of MPS IIIB, as determined by one of the following:

   1. Documented deficiency in alpha-N-acetylglucosaminidase (NAGLU) enzyme activity of ≤10% of the lower limit of the normal range as measured in fibroblasts, leukocytes, plasma, or serum (based on normal range for diagnosis of MPS IIIB). Patients who do not already have a documented deficiency of NAGLU activity will provide a blood sample during screening for determination of NAGLU activity level in their serum. OR
   2. Two documented mutations in the NAGLU gene. Patients who do not already have a documented genotype of NAGLU will provide a blood sample during screening for NAGLU genotyping.
2. The patient is ≥1 and < 10 years of age and has an age equivalent on the Vineland Adaptive Behavior Scales (VABS) of ≥1 year
3. The patient is medically stable, in the opinion of the Investigator, to accommodate the protocol requirements, including travel and assessments, without placing an undue burden on the patient/patient's family.
4. The patient, patient's parent(s) or legal guardian(s) has voluntarily signed and dated an Institutional Review Board/Independent Ethics Committee-approved informed consent (assent if applicable) form after all relevant aspects of the study have been explained and discussed with the patient, the patient's parent(s), or legal guardian(s).Exclusion Criteria:

Patients will be excluded from the study if they meet any of the following criteria at screening:

1. Presence of significant non-MPS IIIB related central nervous system (CNS) impairment or behavioral disturbances, sufficient, in the opinion of the Investigator, to preclude performance of study neurocognitive and developmental testing procedures, or that would confound the scientific integrity or interpretation of study assessments.
2. Visual or hearing impairment sufficient to preclude cooperation with neurodevelopmental testing.
3. Patient has a known or suspected hypersensitivity to anesthesia or is thought to be at an unacceptable risk from anesthesia, due to airway compromise or other conditions, in the opinion of the Investigator.
4. Personal history or family history of neuroleptic malignant syndrome, malignant hyperthermia, or other anesthesia-related concerns.
5. History of poorly controlled seizure disorder.
6. Currently receiving psychotropic or other medications, which in the Investigator's opinion would be likely to substantially confound test results.
7. History of bleeding disorder, inability to abstain from medications that affect blood clotting(e.g., aspirin, Non-steroidal anti-inflammatory drug (NSAIDs)), or history of their ingestion within 1 week prior to a lumbar puncture.
8. History of complications from previous lumbar punctures that, in the opinion of the Investigator, place the patient at increased risk from this procedure.
9. The patient is participating, plans to participate, or participated in a clinical trial of another investigational medicinal product, or has received a vaccination, within the 30 days prior to the study or for less than 5 half lives (whichever is longer) of the investigational product.
10. History of hematopoietic stem cell or bone marrow transplant.
11. Unable to assent, or the patient's parent(s) or patient's legal guardian(s) is/are unable to understand the nature, scope, and possible consequences of the study, or do/does not agree to comply with the protocol defined schedule of assessments.
12. Patient is unable to comply with the protocol (e.g., has a clinically relevant medical condition making implementation of the protocol difficult, unstable social situation, or otherwise unlikely to complete the study) or is, in the opinion of the Investigator, otherwise unsuited for the study.
13. The patient has any item (braces, tattoos, etc) which would exclude the patient from being able to undergo MRI according to local Institutional Policy, or the patient has any other situation that would exclude the patient from undergoing any other procedure required in this study.
14. The patient is pregnant.

Ages: 1 Year to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Patients with a documented diagnosis of MPS IIIB and who are currently untreated with investigational products (drugs/device) for this disease. Patient must also be ≥ 1 year and < 10 years of age with an age equivalent on the Vineland Adaptive Behavior Scales (VABS) of ≥ 1 year.
Sampling Method: Non-Probability Sample
Enrollment: 19 (Actual)
Dates: Start 2012-04-09 (Actual); Primary Completion 2013-10-10 (Actual); Study Completion 2013-10-10 (Actual)

PRIMARY OUTCOMES:
evaluate the course of disease progression in patients with MPS IIIB who are untreated with any investigational products to inform possible future treatment studies | 13 months

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (4):
- United States (2):
  - Children's Hospital and Research Center, Oakland, California
  - University of Minnesota, Minneapolis, Minnesota
- Johannes Gutenberg University Medical Center, Mainz, Germany
- Great Ormond Street Hospital for Children, London, United Kingdom

REFERENCES:
- [Derived] Whitley CB, Cleary M, Eugen Mengel K, Harmatz P, Shapiro E, Nestrasil I, Haslett P, Whiteman D, Alexanderian D. Observational Prospective Natural History of Patients with Sanfilippo Syndrome Type B. J Pediatr. 2018 Jun;197:198-206.e2. doi: 10.1016/j.jpeds.2018.01.044. Epub 2018 Apr 13. PMID 29661560
- See also: To obtain more information on the study, click here/on this link. — https://clinicaltrials.takeda.com/study-detail/5f6b5fcf4db2bf003ab46819